CLINICAL TRIAL: NCT05829785
Title: Influence of Obesity on Microvascular Reactivity During General Anesthesia
Status: Completed | Type: Observational
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Principal Investigator, Hyeon-Jeong Lee, Dr., Pusan National University Hospital
Other Study IDs: 2018-0175; 1804-025-066 (Other: Pusan national university hospital)
Record Dates: First submitted 2023-04-13; First posted 2023-04-26 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Obesity; Anesthesia; Microcirculation
Keywords: Obesity; Body mass index; Anesthesia, general; Microcirculation
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- overweight group: Subjects with a body mass index (BMI) ≥ 25
  Interventions: Device: Near-infrared spectroscopy monitor
- normal weight group: Subjects with BMI < 25
  Interventions: Device: Near-infrared spectroscopy monitor

INTERVENTIONS:
Device: Near-infrared spectroscopy monitor — tissue oxygen saturation monitoring combined with vascular occlusion test

SUMMARY:
The purpose of this study was to investigate the effect of obesity on changes in microvascular reactivity and tissue oxygen saturation (StO2) during general anesthesia using near-infrared spectroscopy in conjunction with vascular occlusion tests (VOT).

For this prospective observation investigation, a total of 128 patients who underwent elective surgery under general anesthesia at Pusan National University Hospital between June 2018 and February 2021 were participated in this study. Baseline StO2 on thenar eminence, hemodynamics, and laboratory profile were monitored before (Tpre) and 30 min after general anesthesia (Tpost). During vascular occlusion tests (VOT), the occlusion slope representing oxygen consumption of muscle and recovery slope representing microvascular reactivity were also collected at Tpre and Tpost. For analysis, the patients were divided into two groups: overweight (body mass index [BMI] ≥ 25 kg/m2) and normal weight (BMI < 25).

DETAILED DESCRIPTION:
Preoperative laboratory findings were obtained. Mean blood pressure (MBP), pulse oxygen saturation (SpO2), heart rate (HR), skin temperature, and VOT-derived measurements, including baseline tissue oxygen saturation (StO2), occlusion slope, minimum StO2, time to minimum StO2, recovery slope, maximum StO2, and time to baseline StO2 were recorded before (Tpre) and 30 min after general anesthesia (Tpost).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who underwent elective surgery under general anesthesia.

Exclusion Criteria:

* Society of Anesthesiologists (ASA) physical status > II
* patients with a neuraxial block
* uncontrolled hypertension
* patients with major cardiovascular disease
* diabetes
* pregnant individuals
* peripheral vascular disease
* chronic venous insufficiency
* smoking: Pack-years > 10
* chronic obstructive and restrictive pulmonary disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who underwent elective surgery under general anesthesia between 2018 and 2021 in Pusan national univ. hospital.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Recovery slope after general aneshtesia (Tpost) | 10 minutes
  Representing microvascular reactivity (Tpost: 30 minutes after general anesthesia); recovery slope was calculated from deflation of the tourniquet until the recovery of StO2 to the baseline value.

SECONDARY OUTCOMES:
Recovery slope before general aneshtesia (Tpre) | 10 minutes
  Representing microvascular reactivity (Tpre: before general anesthesia); recovery slope was calculated from deflation of the tourniquet until the recovery of StO2 to the baseline value.
Occlusion slope before general anesthesia (Tpre) | 10 minutes
  representing oxygen consumption of muscle (Tpre: before general anesthesia); occlusion slope was defined as the slope of StO2 descent to the lowest value.
Occlusion slope before general anesthesia (Tpost) | 10 minutes
  representing oxygen consumption of muscle (Tpost: 30 minutes after general anesthesia); occlusion slope was defined as the slope of StO2 descent to the lowest value.

CONTACTS AND LOCATIONS:
Locations (1):
- Pusan National University Hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cho AR, Lee HJ, Kim HJ, Do W, Jeon S, Baek SH, Kim ES, Kwon JY, Kim HK. Microvascular Reactivity Measured by Dynamic Near-infrared Spectroscopy Following Induction of General Anesthesia in Healthy Patients: Observation of Age-related Change. Int J Med Sci. 2021 Jan 1;18(5):1096-1103. doi: 10.7150/ijms.52433. eCollection 2021. PMID 33526968